CLINICAL TRIAL: NCT02713230
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Study Evaluating the Efficacy, Safety, and Pharmacokinetics of Brachial Plexus Block With EXPAREL for Postsurgical Analgesia in Subjects Undergoing Total Shoulder Arthroplasty or Rotator Cuff Repair
Brief Title: Efficacy, Safety, and Pharmacokinetics of Brachial Plexus Block With EXPAREL in Shoulder Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pacira Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 402-C-327
Record Dates: First submitted 2016-03-15; First posted 2016-03-18 (Estimated); Results first posted 2020-12-03 (Actual); Last update posted 2020-12-03 (Actual); Status verified 2020-11

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- EXPAREL 133 mg (Active Comparator): 10 mL EXPAREL (bupivacaine liposome injectable suspension) expanded with 10 mL normal saline as single-injection brachial plexus block (interscalene or supraclavicular) ≥1 h preoperatively
  Interventions: Drug: bupivacaine liposome injectable suspension
- EXPAREL 266 mg (Active Comparator): 20 mL EXPAREL (bupivacaine liposome injectable suspension) as single-injection brachial plexus block (interscalene or supraclavicular) ≥1 h preoperatively
  Interventions: Drug: bupivacaine liposome injectable suspension
- Placebo (Placebo Comparator): 20 mL normal saline as single-injection brachial plexus block (interscalene or supraclavicular) ≥1 h preoperatively
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: bupivacaine liposome injectable suspension — 10 mL EXPAREL (bupivacaine liposome injectable suspension) expanded with 10 mL normal saline
  Other Names: EXPAREL
  Arms: EXPAREL 133 mg
Drug: bupivacaine liposome injectable suspension — 20 mL EXPAREL (bupivacaine liposome injectable suspension)
  Other Names: EXPAREL
  Arms: EXPAREL 266 mg
Drug: Placebo — 20 mL normal saline as single-injection
  Other Names: Normal saline
  Arms: Placebo

SUMMARY:
This is a Phase 3, multicenter, randomized, double-blind, placebo-controlled study in 155 adult subjects undergoing primary unilateral total shoulder arthroplasty or rotator cuff repair with general anesthesia

DETAILED DESCRIPTION:
On Day 0, eligible subjects will be randomized in a 1:1 ratio to receive a single dose of EXPAREL 133 mg in 10 mL expanded in volume with 10 mL of normal saline for a total volume of 20 mL or placebo 20 mL. Study drug (EXPAREL or placebo) will be administered in a blinded manner via an ultrasound guided single-dose brachial plexus block at least 1 hour prior to surgery.

Postsurgical assessments will include pain intensity scores using a 10-cm visual analog scale (VAS); total postsurgical opioid consumption; overall benefit of analgesia score (OBAS) questionnaire; subject satisfaction with overall analgesia using a 5 point Likert scale; neurological assessment; sensory function assessment; motor function assessment; discharge readiness; unscheduled phone calls or office visits related to pain; 12-lead ECGs; vital sign measurements; and clinical laboratory tests. Adverse events will be recorded from the time the informed consent form is signed through postsurgical Day 29.

Follow-up visits will be scheduled for all subjects on postsurgical Days 5 and 10. A follow-up phone call will be made on postsurgical Day 29.

A population Pharmacokinetic (PK) analysis will be utilized to limit the number of blood draws with a sampling schedule of baseline (prior to the nerve block) through hospital discharge. There will be two collection sequences for this study and a subject can only be randomized to one sequence.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, at least 18 years of age at screening.
2. Scheduled to undergo primary unilateral total shoulder arthroplasty or rotator cuff repair.
3. Subjects scheduled for rotator cuff repair must have a magnetic resonance imaging (MRI) with a reading confirming a tear of at least 1 cm.
4. American Society of Anesthesiologists (ASA) physical status 1, 2, or 3.
5. Female subject must be surgically sterile; or at least 2 years postmenopausal; or have a monogamous partner who is surgically sterile; or practicing double-barrier contraception; or practicing abstinence (must agree to use double-barrier contraception in the event of sexual activity); or using an insertable, injectable, transdermal, or combination oral contraceptive approved by the FDA for greater than 2 months prior to screening and commit to the use of an acceptable form of birth control for the duration of the study and for 30 days after completion of the study.
6. Able to demonstrate normal motor function (by obtaining a 5 on the Lovett Scale when exhibiting biceps, wrist, and thumb movement) and sensory function (by exhibiting sensitivity to cold, pinprick, and light touch) in the location where sensory function will be measured throughout the study: 2 cm superior to the coracoid process on the skin overlying the acromioclavicular joint.
7. Able to provide informed consent, adhere to the study visit schedule, and complete all study assessments.

Exclusion Criteria:

1. Currently pregnant, nursing, or planning to become pregnant during the study or within 1 month after study drug administration.
2. Planned concurrent surgical procedure.
3. Concurrent painful physical condition that may require analgesic treatment (such as an NSAID or opioid) in the postsurgical period for pain that is not strictly related to the shoulder surgery and which may confound the postsurgical assessments (e.g., significant pain from other joints, chronic neuropathic pain).
4. History of hypersensitivity or idiosyncratic reaction to amide-type local anesthetics.
5. Smoking history of greater than 25 pack-years.
6. Contraindication to any one of the following: bupivacaine, oxycodone, morphine, or hydromorphone.
7. Use of any of the following medications within the times specified before surgery: long-acting opioid medications or NSAIDs (except for low-dose aspirin used for cardioprotection) within 3 days, or any opioid medication within 24 hours.
8. Initiation of treatment with any of the following medications within 1 month of study drug administration or if the medication(s) are being given to control pain: selective serotonin reuptake inhibitors (SSRIs), selective norepinephrine reuptake inhibitors (SNRIs), gabapentin, pregabalin (Lyrica®), or duloxetine (Cymbalta®). If a subject is taking one of these medications for a reason other than pain control, he or she must be on a stable dose for at least 1 month prior to study drug administration.
9. Current use of systemic glucocorticosteroids within 1 month of enrollment in this study.
10. Use of dexmedetomidine hydrochloride (HCl) (Precedex®) within 3 days of study drug administration.
11. History of impaired kidney function, emphysema or other chronic respiratory disease, rheumatoid arthritis, coagulopathy, or loss of sensation in extremities.
12. Impaired kidney function (e.g., serum creatinine level >2 mg/dL [176.8 µmol/L] or blood urea nitrogen level >50 mg/dL [17.9 mmol/L]) or impaired liver function (e.g., serum aspartate aminotransferase [AST] level >3 times the upper limit of normal [ULN] or serum alanine aminotransferase [ALT] level >3 times the ULN.)
13. Uncontrolled anxiety, psychiatric, or neurological disorder that might interfere with study assessments.
14. Any chronic neuromuscular deficit effecting the peripheral nerves or muscles of the surgical extremity.
15. Any chronic condition or disease that would compromise neurological or vascular assessments.
16. Malignancy in the last 2 years, with the exception of non-metastatic basal cell or squamous cell carcinoma of the skin or localized carcinoma in situ of the cervix.
17. Suspected or known history of drug or alcohol abuse within the previous year.
18. Body weight <50 kg (110 pounds) or a body mass index >44 kg/m2.
19. Previous participation in an EXPAREL study.
20. Administration of an investigational drug within 30 days or 5 elimination half-lives of such investigational drug, whichever is longer, prior to study drug administration, or planned administration of another investigational product or procedure during the subject's participation in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2016-05-09; Primary Completion 2017-07-07 (Actual); Study Completion 2017-07-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James B Jones, MD, PharmD, Study Director — Pacira Pharmaceuticals, Inc
Locations (20):
- United States (17):
  - Horizon Research Group, Inc, Mobile, Alabama
  - Denver Metro Orthopedics, Englewood, Colorado
  - Jackson Memorial Hospital/University of Miami, Miami, Florida
  - Pensacola Research Associates, Pensacola, Florida
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Montefiore Medical Center, The Bronx, New York
  - Duke University Medical Center, Durham, North Carolina
  - Fairview Hospital, Cleveland, Ohio
  - Indiana Regional Medical Center, Indiana, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Chan Soon-Shiong Medical Center, Windber, Pennsylvania
  - Hermann Drive Surgical Hospital, Houston, Texas
  - Westside Surgical Hospital, Houston, Texas
  - Plano Surgical Hospital, Plano, Texas
  - Houston Physician's Hospital, Webster, Texas
  - Southampton Orthopedics Sports Medicine, Franklin, Virginia
- Ziekenhuis Oost-Limburg, Genk, Belgium
- Denmark (2):
  - Aarhus University Hospital, Aarhus
  - Regionshospital Silkeborg, Silkeborg

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Patel MA, Gadsden JC, Nedeljkovic SS, Bao X, Zeballos JL, Yu V, Ayad SS, Bendtsen TF. Brachial Plexus Block with Liposomal Bupivacaine for Shoulder Surgery Improves Analgesia and Reduces Opioid Consumption: Results from a Multicenter, Randomized, Double-Blind, Controlled Trial. Pain Med. 2020 Feb 1;21(2):387-400. doi: 10.1093/pm/pnz103. PMID 31150095

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited between May 9, 2016 and July 7, 2017 at 16 sites in the US and Europe
Pre-assignment Details: "Started" does not include one patient who was a screen failure, was not enrolled, and was randomized to placebo in error.
Period: Overall Study
Arm/Group | EXPAREL 133 mg | EXPAREL 266 mg | Placebo
Started | 69 | 15 | 71
Completed | 68 | 15 | 71
Not Completed | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety population included all participants who received study drug, with analysis by actual treatment received.
Groups:
- Total: Total of all reporting groups
Arm/Group | EXPAREL 133 mg | EXPAREL 266 mg | Placebo | Total
Number analyzed (Participants) | 69 | 15 | 71 | 155
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.6 (9.94) | 61.4 (7.73) | 58.5 (9.48) | 59.7 (9.55)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 7 | 23 | 55
  Male | 44 | 8 | 48 | 100
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 0 | 5 | 8
  Not Hispanic or Latino | 64 | 15 | 65 | 144
  Unknown or Not Reported | 2 | 0 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 13 | 4 | 15 | 32
  White | 53 | 11 | 54 | 118
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 2 | 4
Region of Enrollment [Count of Participants; unit: Participants]
  Belgium | 7 | 3 | 9 | 19
  United States | 52 | 10 | 53 | 115
  Denmark | 10 | 2 | 9 | 21
Dominant hand [Count of Participants; unit: Participants]
  Left hand | 10 | 1 | 10 | 21
  Right hand | 59 | 14 | 61 | 134
Visual Analog Scale Pain Score [Mean (Standard Deviation); unit: units on a scale] — Visual Analog Scale (VAS) is a pain scale. The VAS was presented as a straight 10 cm line, where 0 cm is no pain and 10 cm is the worst pain possible. Patients were asked, "How much pain are you experiencing right now? Please place a vertical mark on the line below to indicate the level of pain you are experiencing right now."
  units on a scale | 2.43 (2.621) | 2.51 (2.641) | 2.94 (2.514) | 2.68 (2.570)
American Society of Anesthesiologists classification [Count of Participants; unit: Participants] — American Society of Anesthesiologists (ASA) classification was determined by physicians using the ASA Physical Status Classification System which assesses the patient's pre-anesthesia medical co-morbidities. ASA 1 patients would be considered a normal, healthy patient. ASA 2 is a patient with mild systemic disease (eg, smoker, well controlled diabetes or high blood pressure (HBP)). ASA 3 is a patient with severe systemic disease (eg poorly controlled diabetes or HBP). ASA 4 is a patient with severe systemic disease that is a constant threat to life (eg, recent myocardial infarction, stroke).
  Participants
    1 | 15 | 1 | 14 | 30
    2 | 36 | 9 | 37 | 82
    3 | 18 | 5 | 20 | 43
    Greater than or equal to 4 | 0 | 0 | 0 | 0
Type of surgery [Count of Participants; unit: Participants]
  Rotator cuff surgery | 50 | 7 | 55 | 112
  Total shoulder arthroplasty | 19 | 8 | 16 | 43
Nerve block type [Count of Participants; unit: Participants]
  Interscalene | 67 | 15 | 70 | 152
  Supraclavicular | 2 | 0 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Curve (AUC) of Visual Analog Scale (VAS) Pain Intensity Scores
Description: AUC of VAS pain intensity scores through 48 hours, which represents total pain experienced through 48 hours. VAS is a pain scale. The VAS was presented as a straight 10 cm line, where 0 cm is no pain and 10 cm is the worst pain possible. Patients were asked, "How much pain are you experiencing right now? Please place a vertical mark on the line below to indicate the level of pain you are experiencing right now."
Time Frame: 0-48 hours
Population: Efficacy population: all participants who received study drug and underwent the surgery, with analysis based on randomized treatment.
  Under protocol amendment 2, the study arm 266 mg dose of EXPAREL was removed from randomization scheme and efficacy endpoints.
Measure: Least Squares Mean (Standard Error); unit: cm*hr
Arm/Group | EXPAREL 133 mg | Placebo
Number analyzed (Participants) | 69 | 71
cm*hr | 136.431 (12.090) | 254.119 (11.768)
Statistical Analysis 1: Comparison: EXPAREL 133 mg vs Placebo; Test type: Superiority; p < 0.0001, ANOVA; LSMD = -117.688, 95% CI 2-sided [-150.896 to -84.480]

2. Secondary Outcome: Total Postsurgical Opioid Consumption Through 48 Hours
Description: Total postsurgical opioid consumption (converted to IV morphine equivalents) through 48 hours
Time Frame: 0-48 hours
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mg
Arm/Group | EXPAREL 133 mg | Placebo
Number analyzed (Participants) | 69 | 71
mg | 11.973 (2.265) | 54.303 (10.053)
Statistical Analysis 1: Comparison: EXPAREL 133 mg vs Placebo; Test type: Superiority; p < 0.0001, ANOVA; LSM treatment ratio = 0.220, 95% CI 2-sided [0.131 to 0.371]

3. Secondary Outcome: Percentage of Opioid-free Participants Through 48 Hours
Description: Percentage of participants who did not receive opioid medication through 48 hours
Time Frame: 0-48 hours
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | EXPAREL 133 mg | Placebo
Number analyzed (Participants) | 69 | 71
Participants | 9 | 1
Statistical Analysis 1: Comparison: EXPAREL 133 mg vs Placebo; Test type: Superiority; p = 0.008, Cochran-Mantel-Haenszel; Treatment difference = 0.116, 95% CI 2-sided [0.032 to 0.200]

4. Secondary Outcome: Time to First Opioid Rescue Through 48 Hours
Description: Time to first opioid rescue medication consumed through 48 hours. Time to rescue was estimated from Kaplan-Meier analysis and presented as quartiles (ie, time to rescue for the first 25% / 50% / 75% of subjects within each treatment group).
Time Frame: 0-48 hours
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: hours
Arm/Group | EXPAREL 133 mg | Placebo
Number analyzed (Participants) | 69 | 71
hours
  First quartile | 0.70 [0.52 to 1.37] | 0.38 [0.30 to 0.47]
  Median quartile | 4.15 [1.52 to 8.50] | 0.58 [0.48 to 0.68]
  Third quartile | 18.82 [9.73 to 36.40] | 0.87 [0.72 to 1.00]
Statistical Analysis 1: Comparison: EXPAREL 133 mg vs Placebo; Test type: Superiority; p < 0.0001, Log Rank

ADVERSE EVENTS:
Time Frame: From screening to postsurgical day 29
Description: An adverse event (AE) was defined as any untoward medical occurrence associated with the use of a drug in humans whether or not considered drug-related. An AE could therefore have been any unfavorable and unintended sign (eg, abnormal laboratory finding), symptom, or disease temporally associated with the use of a drug without any judgment about causality. Serious AEs were defined as per clinicaltrials.gov.
Arm/Group | EXPAREL 133 mg | EXPAREL 266 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/69 | 0/15 | 0/71
Serious Adverse Events (participants affected / at risk) | 2/69 | 1/15 | 1/71
Other Adverse Events (participants affected / at risk) | 55/69 | 11/15 | 55/71
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | EXPAREL 133 mg (N=69) | EXPAREL 266 mg (N=15) | Placebo (N=71)
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 1 | 0
Gout (Metabolism and nutrition disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | EXPAREL 133 mg (N=69) | EXPAREL 266 mg (N=15) | Placebo (N=71)
Nausea (Gastrointestinal disorders) | 17 | 3 | 26
Constipation (Gastrointestinal disorders) | 6 | 2 | 9
Vomiting (Gastrointestinal disorders) | 4 | 1 | 7
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 4
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0
Dizziness (Nervous system disorders) | 2 | 1 | 9
Headache (Nervous system disorders) | 7 | 1 | 3
Dysgeusia (Nervous system disorders) | 6 | 0 | 3
Hypoesthesia (Nervous system disorders) | 6 | 0 | 1
Paresthesia (Nervous system disorders) | 1 | 1 | 1
Sensory loss (Nervous system disorders) | 2 | 1 | 0
Pyrexia (General disorders) | 6 | 1 | 3
Pruritis (Skin and subcutaneous tissue disorders) | 3 | 1 | 11
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Muscle twitching (Musculoskeletal and connective tissue disorders) | 5 | 2 | 8
Hypertension (Vascular disorders) | 2 | 3 | 6
Hypotension (Vascular disorders) | 1 | 1 | 2
Insomnia (Psychiatric disorders) | 2 | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 1 | 0
Tachycardia (Cardiac disorders) | 1 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Results conducted at Site shall not be published before 1st multicenter publication by Sponsor but can proceed if there is no such publication ≤18 months after study completion/termination at all sites and all data have been received. Before submitting manuscript/materials to an outside person/entity, site shall give Sponsor 60 days to review and comment. Site shall, upon request, further delay publication/presentation for ≤120 days to allow Sponsor to protect its interests in Inventions.

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-06-26): https://cdn.clinicaltrials.gov/large-docs/30/NCT02713230/SAP_000.pdf
  • Study Protocol (2016-11-14): https://cdn.clinicaltrials.gov/large-docs/30/NCT02713230/Prot_001.pdf